CLINICAL TRIAL: NCT04171037
Title: A Pilot Study of FDA Approved Optiflow™ THRIVE Versus Standard Non-Rebreathers in Patients With Potential High Risk of Airway Obstruction During Total Intravenous Anesthesia (TIVA) While Undergoing Interventional Radiology Procedures
Brief Title: Optiflow THRIVE for Delivery of Oxygen to Patients During Total Intravenous Anesthesia While Undergoing Radiology Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-0348; NCI-2019-07291 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0348 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-11-19; First posted 2019-11-20 (Actual); Results first posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm I (oxygen via Optiflow THRIVE) (Experimental): Patients receive 100% oxygen at a high flow rate via Optiflow THRIVE over 3 minutes prior to anesthetic induction and at a higher flow rate until the end of procedure.
  Interventions: Procedure: Oxygen Therapy; Other: Questionnaire Administration; Device: Optiflow THRIVE
- Arm II (oxygen via non-rebreather mask) (Active Comparator): Patients receive 100% oxygen at a lower flow rate via non-rebreather mask over 3 minutes prior to anesthetic induction and maintain the same flow rate until the end of procedure.
  Interventions: Procedure: Oxygen Therapy; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Oxygen Therapy — Receive oxygen via Optiflow THRIVE
  Other Names: supplemental oxygen therapy
  Arms: Arm I (oxygen via Optiflow THRIVE)
Procedure: Oxygen Therapy — Receive oxygen via non-rebreather
  Other Names: supplemental oxygen therapy
  Arms: Arm II (oxygen via non-rebreather mask)
Other: Questionnaire Administration — Ancillary studies
Device: Optiflow THRIVE — Oxygen Administration
  Arms: Arm I (oxygen via Optiflow THRIVE)

SUMMARY:
This trial studies how well Optiflow THRIVE works in delivering oxygen to patients during total intravenous anesthesia while undergoing radiology procedures. The Optiflow THRIVE is an oxygen administration device that delivers high-flow and humidified oxygen through the nose. The Optiflow THRIVE device may improve oxygen delivery and reduce breathing complications.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To investigate the performance of Optiflow THRIVE relative to Standard Non-Rebreathers in patients with high risk of difficult airway management undergoing interventional radiology procedures for the planning of future clinical studies.

SECONDARY OBJECTIVE:

I. To describe the episodes of hypoxia (defined by peripheral capillary oxygen saturation [SpO2] less than or equal to 92%) and the episodes of airway support which include: jaw thrust, chin lift or insertion of an airway supporting device, such as oral/nasal airway or supra airway device in order to recover the level of oxygenation above 92% associated with Optiflow THRIVE.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive 100% oxygen at a high flow rate via Optiflow THRIVE over 3 minutes prior to anesthetic induction and at a higher flow rate until the end of procedure.

ARM II: Patients receive 100% oxygen at a lower flow rate via non-rebreather mask over 3 minutes prior to anesthetic induction and maintain the same flow rate until the end of procedure.

After completion of study, patients are followed up at 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent for the study
* Patients with an SpO2 greater than or equal to 95% while breathing room air
* Patients requiring total intravenous anesthesia (TIVA) but not tracheal intubation during the proposed procedure - PLUS, any of the 2 following criteria: Body mass index (BMI) greater than or equal to 32 kg/m^2, or neck circumference greater than or equal to 43 cm in a male and 41 cm in a female, or has been diagnosed with moderate to severe obstructive sleep apnea (OSA) with/without using a continuous positive airway pressure (CPAP) device
* Full course head and neck radiotherapy less than or equal to 6 months (the peak onset time of acute facial and airway edema)

Exclusion Criteria:

* Significant pulmonary disease requiring supplemental oxygen in daily life (severe pulmonary fibrosis, severe chronic obstructive pulmonary disease, etc.)
* Significant cardiac disease (including history of myocardial infarction [MI] with concurrent evidence of ischemic myocardial damage at the event, cardiomyopathy with impaired left ventricular ejection fraction to less than 50% or uncompensated congestive heart failure)
* TIVA is contraindicate or having a proposed procedure without TIVA
* Endotracheal intubation is required
* American Society of Anesthesiologists (ASA) physical status classification 5
* Patients who are non-English speaking
* Emergency procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gang Zheng, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The IR procedure daily schedule will be used for patient selection. Once eligibility of a study candidate has been identified, the study coordinator will be informed to start the patient interview and obtain written informed consent.
Pre-assignment Details: A total of 114 patients were accrued, and 108 patients were randomized. Of the total number randomized, six patients were screen failures prior to the procedure and 1 patient had no follow-up measurements, leaving 101 patients deemed evaluable for the primary endpoint. This provided 50 patients on Optiflow THRIVE and 51 patients on Standard of Care.
Groups:
- Optiflow™ THRIVE: Treatment group will receive oxygen via Optiflow™ THRIVE
- Control Group (Non-rebreather Facemask): Control group will receive 100% oxygen via a non-rebreather facemask
Period: Overall Study
Arm/Group | Optiflow™ THRIVE | Control Group (Non-rebreather Facemask)
Started | 54 | 54
Completed | 50 | 51
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Optiflow™ THRIVE | Control Group (Non-rebreather Facemask) | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 32 | 62
  >=65 years | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.18 (11.96) | 60.96 (11.97) | 60.57 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 28 | 28 | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 50 | 51 | 101

OUTCOME MEASURES:

1. Primary Outcome: Total Length of Desaturation Episodes (ToLDE) Per Patient/Surgical Procedure
Description: This measure is defined as the total length (in minutes) of all desaturation episodes that a patient experienced during a 60-minute observation window starting from the initiation of the propofol infusion. A desaturation episode is defined as a drop in oxygen saturation (SpO2) to 92% or lower.
Time Frame: 60-minute observation window starting from the initiation of the propofol infusion and continuing for 60 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Optiflow™ THRIVE | Control Group (Non-rebreather Facemask)
Number analyzed (Participants) | 50 | 51
minutes | 34 (1.16) | 97 (3.25)

2. Secondary Outcome: Number of Desaturation Episode Events Per Patient/Surgical Procedure
Description: The total number of episodes where the patient's oxygen saturation (SpO2) dropped to 92% or lower.
Time Frame: 60-minute observation window starting from the initiation of the propofol infusion and continuing for 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Optiflow™ THRIVE | Control Group (Non-rebreather Facemask)
Number analyzed (Participants) | 50 | 51
Participants | 7 | 13

3. Secondary Outcome: Number of BIS Episodes
Description: The total number of episodes where the bispectral index (BIS) value was 61 or higher, indicating inadequate sedation levels.
Time Frame: 60-minute observation window starting from the initiation of the propofol infusion.
Measure: Median (Full Range); unit: Number of Episodes
Arm/Group | Optiflow™ THRIVE | Control Group (Non-rebreather Facemask)
Number analyzed (Participants) | 50 | 51
Number of Episodes | 2 [0 to 15] | 4 [0 to 19]

4. Secondary Outcome: PACU Observation Time
Description: The length of time spent in the post-anesthesia care unit (PACU) in minutes.
Time Frame: up to 60 minutes after PACU admission
Measure: Median (Full Range); unit: minutes
Arm/Group | Optiflow™ THRIVE | Control Group (Non-rebreather Facemask)
Number analyzed (Participants) | 50 | 51
minutes | 20 [0 to 60] | 26 [0 to 60]

ADVERSE EVENTS:
Time Frame: From Induction to 15 minutes after PACU arrival
Arm/Group | Optiflow™ THRIVE | Control Group (Non-rebreather Facemask)
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/51
Other Adverse Events (participants affected / at risk) | 0/50 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT04171037/Prot_SAP_000.pdf